CLINICAL TRIAL: NCT01116050
Title: Second-line Treatment of Post-partum Haemorrhage With Intrarectal Misoprostol: a Multicentre, Double Blind, Randomized Placebo-controlled Trial
Brief Title: Intrarectal Misoprostol in Postpartum Haemorrhage
Acronym: HEMOSTOP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Monsieur Angel PIQUEMAL, Caen University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03-104; 03-104
Record Dates: First submitted 2010-05-03; First posted 2010-05-04 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-05

CONDITIONS: Postpartum Haemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- MISOPROSTOL (Experimental)
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — 5 tablets of 200 microgram geach intra rectal by opaque introducer
  Arms: MISOPROSTOL
Drug: Placebo — 5 tablets in opque introducer
  Arms: Placebo

SUMMARY:
Postpartum haemorrhage (PPH) remains the major cause of maternal mortality in France. The most efficient treatment of severe PPH is sulprostone which is associated with cardiac complications. The objective of this study was to assess the efficacy and the safety of intrarectal misoprostol for curative postpartum haemorrhage treatment.

We conducted a multicenter double blind randomized placebo control trial between June 2004 and December 2007, among consenting women with postpartum haemorrhage and failure to oxytocin treatment.

Our main criteria of judgement was quantification of blood loss and the use of sulprostone between the two groups using either misoprostol intrarectal tablets (5X200mg ) or placebo in similar opaque introducer.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 yrs old
* Giving birth after 32 Weeks of amenorrhea
* Post-partum haemorrhage due to atony
* Inefficiency off the first line treatment
* Written signed consent form

Exclusion Criteria:

* known allergy to prostaglandin
* haemostasis anomalies before labour
* anticoagulant treatment
* fetal death
* accreta or percreta placenta
* under 18 years
* delivery before 32 weeks of amenorrhea
* post-partum bleeding not suspected to be due to atonic uterus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2004-01; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
quantification of blood loss | 15 minutes after treatment administration
  quantification of blood loss and the use of sulprostone between the two groups using either misoprostol intrarectal tablets (5X200mg ) or placebo in similar opaque introducer

SECONDARY OUTCOMES:
Sulprostone Requirement | 30 minutes after the diagnostic of post-partum hemorrhage
  distribution of blood loss over time, blood loss higher than 500mL after treatment, blood transfusion, changes in haemoglobin concentration and haematocrit levels, recourse to sulprostone, uterine arteries embolizations and hysterectomy

CONTACTS AND LOCATIONS:
Overall Officials: Michel DREYFUS, MD, PhD, Principal Investigator — University Hospital, Caen

REFERENCES:
- [Derived] Parry Smith WR, Papadopoulou A, Thomas E, Tobias A, Price MJ, Meher S, Alfirevic Z, Weeks AD, Hofmeyr GJ, Gulmezoglu AM, Widmer M, Oladapo OT, Vogel JP, Althabe F, Coomarasamy A, Gallos ID. Uterotonic agents for first-line treatment of postpartum haemorrhage: a network meta-analysis. Cochrane Database Syst Rev. 2020 Nov 24;11(11):CD012754. doi: 10.1002/14651858.CD012754.pub2. PMID 33232518